CLINICAL TRIAL: NCT04678700
Title: Implementation of a Respiratory Physiotherapy Program in Post COVID-19 Patients Through Tele-assistance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: European University of Madrid (Other)
Responsible Party: Principal Investigator, Marta de la Plaza, Physiotherapy teacher, PH student, European University of Madrid
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20/139
Record Dates: First submitted 2020-12-12; First posted 2020-12-22 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2020-12

CONDITIONS: Covid19- Coronavirus- Sars-cov-2
Keywords: chest physiotherapy; covid19; pulmonary rehabilitation covid19; physical therapy; coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Intervention Model Description: Experimental study composed of an intervention group and a control group The control group will receive the intervention after finishing the intervention with the experimental group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental groupe (Experimental): Intervention; 10 sessions telematics. Before starting and at the end of the respiratory physiotherapy program, the patient complete an online form which includes a quality of life questionnaire, an effort dyspnea questionnaire and an anxiety questionnaire.
  The intervention of the following study follow the recommendations of chest physiotherapy in the management of the patient post covid-19 (1)(17).
  Pre-session; respiratory frequency, dyspnea, oxigenation level are taken. Breathing techniques;
  * Abdominal-diaphragmatic breathing(1)(16). (10 times).
  * Costal expansion exercises with flexion and abduction of the upper limbs. (10 times)(1).
  * Self-passive stretching of the ribcage and neck muscles, accessory to inspiration(25)(26).
  * Jacobson's progressive relaxation(27). Post-session, respiratory frequency and the Borg's dyspnea index/ oxigenation level.
  Interventions: Other: Chest physiotherapy post-covid19
- control groupe (Other): The control group will complete the same questionnaires before and after the intervention, which will give us an idea of whether our intervention has had any improvement. In order for all patients to be able to receive the therapy if they want to. The control group will be on the waiting list to perform the sessions.
  Interventions: Other: Chest physiotherapy post-covid19

INTERVENTIONS:
Other: Chest physiotherapy post-covid19 — The sessions are divided into the following modules;
  * Directed abdominal-diaphragmatic ventilation (10 times).
  * Costal expansion exercises with the help of flexion and abduction of the upper limbs. (10 times)(1).
  * Self-passive stretching of the ribcage and neck muscles, accessory to inspiration. The purpose of the stretching will be to increase the flexibility of the muscles to improve the vital capacity as has already been evidenced in other respiratory diseases such as chronic obstructive pulmonary disease (COPD) and cystic fibrosis (25)(26).
  Relaxation time;Jacobson's progressive relaxation; we scan the body's condition.
  Post-session evaluation by taking the respiratory frequency/ min and the Borg's dyspnea index, and level oxigen after the exercises.

SUMMARY:
The objective of this research project is to scientifically evidence a pulmonary rehabilitation program that was initiated altruistically during the confinement of those patients who had suffered from COVID-19, through an online platform.

Patients are connected telematically 3 times a week from April 6, 2020 to perform the physical therapy program. Due to the clinical improvements that have been referred by patients, they began to take objective data.

Our goal is to know if a telematic respiratory therapy program in post-covid 19 patient, improves the level of anxiety, dyspnea on effort, improves quality of life and oxygenation.

DETAILED DESCRIPTION:
Patients affected by COVID- 19 have long periods of convalescence at home. This fact, together with the measures of social isolation, has contributed to act from a new therapeutic paradigm with the implementation of telematic rehabilitation programs.

On April 6, 2020 the online platform was born under the name "Respiratory Physiotherapy; telematic assistance in patients with COVID-19 sequelae".

We want to quantify the Chest Physiotherapy online program.

Hypothesis; An online respiratory physiotherapy program offers improvements in quality of life, dyspnea and anxiety to patients who have suffered COVID-19.

Objectives; General objective; To improve the pulmonary function of patients who have suffered from COVID-19 infection through an online respiratory physiotherapy program.

Secondary objectives;

* To improve the sensation of dyspnea; quantified by the Malher and Borg scale
* To Normalize Breathing Rate
* To Improve oxigenation; pulse-oximetry
* To Improve the quality of life; quantified Euroqol- 5D
* To Improve the feeling of anxiety; quantified by the STAI questionnaire

METHODOLOGY/STUDY DESIGN; This is a program that was born under a very special need and circumstance, as is the coronavirus pandemic. The aim was to use respiratory tele-rehabilitation through an online platform with patients affected by coronavirus.

The study is voluntary, the patient can stop the program at any time he or she considers appropriate. All of this is informed in the consent form that you give us, duly signed.

I

ELIGIBILITY:
Inclusion Criteria:

* Patients in the recovery phase, hospitalised or at home.
* Patients diagnosed with positive PCR for COVID-19
* Patient with sensation of dyspnea
* Patient able to sit still

Exclusion Criteria:

* Patients admitted to intensive care and/or hemodynamically unstable
* Patients connected to mechanical ventilation
* Patients who do not have integrated cognitive abilities
* Patients who are receiving other respiratory rehabilitation programs
* Patients without adecuate technologies ( WIFI, computer, email, zoom)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Euroqol-5d european quality of life-5 dimensions | 1 week
  The EQ-5D is a generic Quality of Life measurement instrument. The individual himself evaluates his state of health, first in levels of severity by dimensions. The descriptive system contains five health dimensions (mobility, self-care, activities of daily living, pain/discomfort and anxiety/depression) and each one has three levels of severity (no problems, some moderate problems or problems and serious problems). In this part of the questionnaire, the individual must mark the level of severity corresponding to his or her state of health in each one of the dimensions, referring to the same day that he or she completes the questionnaire. In each dimension of the EQ-5D, the levels of severity are coded with a 1 if the answer option is "no (I have) problems"; with a 2 if the answer option is "some or moderate problems"; and with a 3 if the answer option is "many problems".
Euroqol-5d european quality of life-5 dimensions | 4 week
  The EQ-5D is a generic Quality of Life measurement instrument. The individual himself evaluates his state of health, first in levels of severity by dimensions. The descriptive system contains five health dimensions (mobility, self-care, activities of daily living, pain/discomfort and anxiety/depression) and each one has three levels of severity (no problems, some moderate problems or problems and serious problems). In this part of the questionnaire, the individual must mark the level of severity corresponding to his or her state of health in each one of the dimensions, referring to the same day that he or she completes the questionnaire. In each dimension of the EQ-5D, the levels of severity are coded with a 1 if the answer option is "no (I have) problems"; with a 2 if the answer option is "some or moderate problems"; and with a 3 if the answer option is "many problems".
Dysnea scale Borg | 5 minutes before each session
  The modified Borg scale is a visual analog scale standardized in Spanish that allows to evaluate the subjective perception of the breathing difficulty or the physical effort exercised.
  This variable is taken in sedation
Dysnea scale Borg | 5 minutes after each session
  The modified Borg scale is a visual analog scale standardized in Spanish that allows to evaluate the subjective perception of the breathing difficulty or the physical effort exercised.
  This variable is taken in sedation
Respiratory rate | 5 minutes before each session
  breathing rate in one minute. The patient sitting upright takes the number of breaths per minute.
Respiratory rate | 5 minutes after each session
  breathing rate in one minute. The patient sitting upright takes the number of breaths per minute.
Effort dysnea Scale | 1 week
  Effort dyspnea scale, Malher Scale A multidimensional scale that measures 3 magnitudes of dyspnea at a given time: the difficulty of the task, the intensity of the effort and the functional impairment.
Effort dysnea Scale | 4 week
  Effort dyspnea scale, Malher Scale A multidimensional scale that measures 3 magnitudes of dyspnea at a given time: the difficulty of the task, the intensity of the effort and the functional impairment.
Anxiety | 1 week
  STAI, questionary of anxiety, we will take before the first session and at the end of the last session
Anxiety | 4 week
  STAI, questionary of anxiety, we will take before the first session and at the end of the last session
Level oxigen % | 1 week
  pulxe-oximetry, the patient is sitting at rest
Level oxigen % | 4 week
  pulxe-oximetry, the patient is sitting at rest

CONTACTS AND LOCATIONS:
Overall Officials: Marta de la plaza, Principal Investigator — European University of Madrid
Locations (1):
- Marta de la plaza, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No